CLINICAL TRIAL: NCT04700124
Title: A Phase 3, Randomized, Open-label Study to Evaluate Perioperative Enfortumab Vedotin Plus Pembrolizumab (MK-3475) Versus Neoadjuvant Gemcitabine and Cisplatin in Cisplatin-eligible Participants With Muscle-invasive Bladder Cancer (KEYNOTE-B15 / EV-304)
Brief Title: Perioperative Enfortumab Vedotin (EV) Plus Pembrolizumab (MK-3475) Versus Neoadjuvant Chemotherapy for Cisplatin-Eligible Muscle Invasive Bladder Cancer (MIBC) (MK-3475-B15/ KEYNOTE-B15 / EV-304)
Acronym: KEYNOTE-B15
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: Seagen Inc. (Industry); Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3475-B15; MK-3475-B15 (Other: MSD); KEYNOTE-B15 (Other: MSD); EV-304 (Other: MSD); jRCT2041210011 (Registry Identifier: jRCT); PHRR221021-005086 (Registry Identifier: Philippine Health Research Registry (PHRR)); 2023-505615-21-00 (Registry Identifier: EU CT); U1111-1292-1300 (Registry Identifier: UTN); 2020-003106-31 (EudraCT Number)
Record Dates: First submitted 2021-01-05; First posted 2021-01-07 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Bladder Cancer
Keywords: Programmed cell death 1 (PD-1); Programmed Death-Ligand 1 (PD-L1); Programmed Death-Ligand 2 (PD-L2); Pelvic Lymph Node Dissection (PLND); Radical Cystectomy (RC)
MeSH Terms: conditions — Urinary Bladder Neoplasms; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab; enfortumab vedotin; Surgical Procedures, Operative; Gemcitabine; Cisplatin

STUDY DESIGN:
Masking Description: Open label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A: Perioperative EV+ Pembrolizumab and RC + PLND (Experimental): Participants receive 4 cycles (each cycle length = 21 days) of EV intravenous (IV) infusion plus pembrolizumab IV infusion preoperatively, followed by RC + PLND, followed by 5 cycles of adjuvant EV IV infusion plus 13 cycles of adjuvant pembrolizumab IV infusion postoperatively. The total treatment duration is up to approximately 1 year.
  Interventions: Biological: Pembrolizumab; Biological: Enfortumab vedotin (EV); Procedure: RC + PLND
- Arm B: Standard of Care (SOC)-Neoadjuvant chemotherapy (gemcitabine + cisplatin) and RC + PLND (Active Comparator): Participants receive 4 cycles (each cycle length = 21 days) of standard of care (SOC) chemotherapy (gemcitabine IV infusion plus cisplatin IV infusion) preoperatively, followed by RC + PLND. The total treatment duration is up to approximately 3 months.
  Interventions: Procedure: RC + PLND; Drug: Gemcitabine; Drug: Cisplatin

INTERVENTIONS:
Biological: Pembrolizumab — 200 mg of Pembrolizumab IV infusion, on Day 1 Q3W for 4 cycles (each cycle length = 21 days) in preoperative phase (up to approximately 3 months) and on Day 1 Q3W for 13 cycles in postoperative phase (up to approximately 9 months). The total duration of treatment is up to approximately 1 year.
  Other Names: KEYTRUDA®; MK-3475
  Arms: Arm A: Perioperative EV+ Pembrolizumab and RC + PLND
Biological: Enfortumab vedotin (EV) — 1.25 mg/kg of EV IV infusion, on Day 1 and Day 8 Q3W for 4 cycles (each cycle length = 21 days) in preoperative phase (up to approximately 3 months) and on Day 1 and Day 8 Q3W for 5 cycles (each cycle length = 21 days) in postoperative phase (up to approximately 4 months). The total duration of treatment is up to approximately 7 months.
  Other Names: Padcev
  Arms: Arm A: Perioperative EV+ Pembrolizumab and RC + PLND
Procedure: RC + PLND — Curative intent RC + PLND surgery will be administered to all participants randomized to Arm A and B after completion of preoperative systemic treatment (RC + PLND to be done approximately at 15 weeks from randomization).
  Other Names: Surgery
Drug: Gemcitabine — 1000 mg/m^2 of Gemcitabine IV infusion, Day 1 and Day 8 Q3W for 4 cycles in preoperative phase (up to approximately 3 months)
  Other Names: Gemzar
  Arms: Arm B: Standard of Care (SOC)-Neoadjuvant chemotherapy (gemcitabine + cisplatin) and RC + PLND
Drug: Cisplatin — 70 mg/m^2 of Cisplatin IV infusion, Day 1, Q3W for 4 cycles in preoperative phase (up to approximately 3 months)
  Other Names: Platinol®; Platinol®-AQ
  Arms: Arm B: Standard of Care (SOC)-Neoadjuvant chemotherapy (gemcitabine + cisplatin) and RC + PLND

SUMMARY:
The purpose of this study is to assess the antitumor efficacy and safety of perioperative enfortumab vedotin (EV) plus pembrolizumab and radical cystectomy (RC) + pelvic lymph node dissection (PLND) compared with the current standard of care (neoadjuvant chemotherapy [gemcitabine plus cisplatin] and RC + PLND) for participants with MIBC who are cisplatin-eligible. The primary hypothesis is perioperative EV and pembrolizumab and RC + PLND (Arm A) will achieve superior event free survival (EFS) compared with neoadjuvant gemcitabine + cisplatin and RC + PLND (Arm B).

ELIGIBILITY:
Inclusion Criteria:

* Have a histologically confirmed diagnosis of urothelial carcinoma (UC) / muscle invasive bladder cancer (MIBC) (T2-T4aN0M0 or T1-T4aN1M0) with predominant (≥50%) urothelial histology.
* Have clinically non-metastatic bladder cancer (N≤1 M0) determined by imaging (computed tomography (CT) or magnetic resonance imaging (MRI) of the chest/abdomen/pelvis
* Be deemed eligible for Radical Cystectomy (RC) + Pelvic Lymph Node Dissection (PLND)
* Have Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Have adequate organ function.

Exclusion Criteria:

* Has a known additional malignancy that is progressing or has required active anti-cancer treatment ≤3 years of study randomization with certain exceptions
* Has received any prior systemic treatment for MIBC or non-invasive muscle bladder cancer (NMIBC - prior treatment for NMIBC with intravesical BCG/chemotherapy is permitted) or prior therapy with an anti- programmed cell death 1 (PD-1), anti-programmed cell death ligand 1/ ligand 2 (PD-L1/L2), or anti-cytotoxic T-lymphocyte-associated protein 4 (CTLA-4)
* Has ≥N2 disease or metastatic disease (M1) as identified by imaging
* Is cisplatin-ineligible, as defined by meeting any one of the cisplatin ineligibility criteria as per protocol
* Has received prior systemic anticancer therapy including investigational agents within 3 years of randomization or any radiotherapy to the bladder
* Has undergone partial cystectomy of the bladder to remove any NMIBC or MIBC
* Has received a live or live attenuated vaccine within 30 days before the first dose of study intervention
* Has a diagnosis of immunodeficiency or has a known history of human immunodeficiency virus (HIV) infection. Hepatitis B infection or known active Hepatitis C infection
* Has a known psychiatric or substance abuse disorder
* Has had an allogenic tissue/solid organ transplant
* Has ongoing sensory or motor neuropathy Grade 2 or higher
* Has active keratitis (superficial punctate keratitis) or corneal ulcerations
* Has a history of uncontrolled diabetes defined as hemoglobin A1c (HbA1c) ≥8% or HbA1c 7% to <8% with associated diabetes symptoms

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 808 (Actual)
Dates: Start 2021-04-21 (Actual); Primary Completion 2025-10-27 (Actual); Study Completion 2025-10-27 (Actual)

PRIMARY OUTCOMES:
Event-Free Survival (EFS) | Up to ~68 months
  EFS is defined as the time from randomization to the first occurrence of following events: radiographic disease progression precluding RC + PLND, failure to undergo surgery in participants with residual disease, gross residual disease left behind at time of surgery, local or distant recurrence based on blinded independent central review (BICR) or death due to any cause.

SECONDARY OUTCOMES:
Pathologic Complete Response (pCR) Rate | Up to ~47 months
  pCR rate is defined as defined as the proportion of participants having pCR. pCR is defined as absence of viable tumor (pT0N0) in examined tissue from radical cystectomy (RC) + pelvic lymph node dissection (PLND), as assessed by blinded central pathologic review.
Overall Survival (OS) | Up to ~68 months
  OS is defined as the time from randomization to death due to any cause.
Disease Free Survival (DFS) | From ~12 months to up to ~68 months
  DFS is defined as the time from postsurgery baseline scan until the first occurrence of either local/distant recurrence as assessed by BICR imaging and/or biopsy or death from any cause.
Pathologic Downstaging (pDS) Rate | Up to ~47 months
  pDS is defined as participants with <pT2 (includes pT0, pTis, pTa, and pT1) and N0 in examined tissue from RC plus PLND, based on central pathologic review.
Number of Participants Who Experienced An Adverse Event (AE) (Arm A only) | Up to ~68 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants who experience an AE will be presented.
Number of Participants Who Discontinued Study Treatment Due to An AE (Arm A only) | Up to ~68 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants who discontinue study treatment due to an AE will be presented.
Number of Participants Experiencing Perioperative Complications | Up to ~68 months
  Perioperative complications are defined as both intraoperative and postoperative complications, potentially contributing to increased length of inpatient care and/or delay of adjuvant therapy. The number of participants experiencing perioperative complications will be presented.
Change from Baseline in the European Organization for Research and Treatment of Cancer (EORTC)-Quality of Life Questionnaire-Core 30 (QLQ-C30) Global Health Status/Quality of Life (Items 29 and 30) Combined Score | Baseline, Up to ~68 months
  The EORTC QLQ-C30 is a 30-item questionnaire to assess the overall quality of life in cancer participants. Participant responses to questions 29 ("How would you rate your overall health during the past week?") and 30 ("How would you rate your overall quality of life during the past week?") are scored on a 7-point scale (1= Very poor to 7=Excellent). A higher score indicates a better overall health/quality of life status. The change from baseline in EORTC QLQ-C30 Items 29 and 30 combined scores will be presented.
Change from Baseline in EORTC QLQ-C30 Physical Functioning Scale | Baseline, Up to ~68 months
  The EORTC QLQ-C30 is a 30-item questionnaire to assess the overall quality of life of cancer patients. Participant responses to 5 questions about their physical functioning are scored on a 4-point scale (1=not at all to 4=very much). A higher score indicates a better quality of life. The change from baseline in physical function (EORTC QLQ-C30 Items 1-5) score will be presented.
Change From Baseline in Urinary, Bowel and Sexual Domains per Bladder Cancer Index (BCI) | Baseline, Up to ~68 months
  The BCI is a 36-item validated, condition-specific health questionnaire to assess the quality of life among participants with bladder cancer. The BCI contains 3 domains: urinary (14 items), bowel (10 items), and sexual (12 items) with function (Likert response scale: 0 [Never] - 4 [Always]) and bother (Likert response scale: 0 [No problem] - 4 [Big problem]) subdomains. The domain and subdomain scores are standardized to a 0 to 100 point scale where higher scores correspond better functioning and health-related qualify of life. The change from baseline in the combined scores of the urinary, bowel, and sexual domains of the BCI will be presented.
Change from Baseline in EuroQoL-5 Dimensions, 5-level Questionnaire (EQ-5D-5L) Visual Analogue Score (VAS) | Baseline, Up to ~68 months
  The EQ-5D-5L VAS records the respondent's self-rated health on a 10 centimeter (cm) vertical, visual analogue scale. It is rated by the respondent on a scale 0 to 100, with 0 being "the worst health you can imagine" and 100 being "the best health you can imagine". The change from baseline in EQ-5D-5L VAS will be presented.
Change from Baseline in EORTC QLQ-C30 Role Functioning Combined Score (Items 6-7) | Baseline, Up to ~68 months
  The EORTC QLQ-C30 is a 30-item questionnaire to assess the overall quality of life of cancer patients. Participant responses to the questions "Were you limited in doing either your work or other daily activities during the past week?" and " Were you limited in pursuing your hobbies or other leisure time activities during the past week?" will be scored on a 4-point scale (1=Not at All to 4=Very Much). Higher scores indicate a better level of role functioning. Change from baseline in the role functioning (EORTC QLQ-C30 Items 6-7) combined score will be presented.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (188):
- United States (22):
  - Mayo Clinic in Arizona - Phoenix ( Site 0043), Phoenix, Arizona
  - St Joseph Heritage Healthcare-Oncology ( Site 0035), Fullerton, California
  - UCLA Hematology/Oncology - Westwood (Building 200 Suite 140)-Department of Urology/Institute of Uro ( Site 0005), Los Angeles, California
  - University of California San Francisco ( Site 0010), San Francisco, California
  - Stanford University ( Site 0023), Stanford, California
  - University of Colorado, Anschutz Cancer Pavilion ( Site 0009), Aurora, Colorado
  - UF Health ( Site 0031), Gainesville, Florida
  - Indiana University Melvin and Bren Simon Cancer Center ( Site 0050), Indianapolis, Indiana
  - University of Iowa Hospital and Clinics ( Site 0029), Iowa City, Iowa
  - University of Louisville, James Graham Brown Cancer Center ( Site 0022), Louisville, Kentucky
  - Icahn School of Medicine at Mount Sinai ( Site 0011), New York, New York
  - White Plains Hospital ( Site 0039), White Plains, New York
  - Duke University Medical Center ( Site 0017), Durham, North Carolina
  - Wake Forest Baptist Health ( Site 0014), Winston-Salem, North Carolina
  - Oregon Health and Science University ( Site 0028), Portland, Oregon
  - MidLantic Urology ( Site 0002), Bala-Cynwyd, Pennsylvania
  - Saint Francis Cancer Center ( Site 0008), Greenville, South Carolina
  - The University of Tennessee Medical Center ( Site 0034), Knoxville, Tennessee
  - UT Southwestern Medical Center ( Site 0003), Dallas, Texas
  - Houston Methodist Urology Associates ( Site 0033), Houston, Texas
  - Urology of San Antonio ( Site 0020), San Antonio, Texas
  - University of Wisconsin Hospital and Clinics ( Site 0037), Madison, Wisconsin
- Argentina (6):
  - Hospital Británico de Buenos Aires-Oncology ( Site 1551), Ciudad Autónoma de Buenos Aires, Buenos Aires
  - Hospital Italiano de Buenos Aires ( Site 1554), ABB, Buenos Aires F.D.
  - Asociación de Beneficencia Hospital Sirio Libanés ( Site 1553), Buenos Aires, Buenos Aires F.D.
  - Centro de Educación Médica e Investigaciones Clínicas (CEMIC) ( Site 1558), Buenos Aires, Buenos Aires F.D.
  - Fundacion Estudios Clinicos-Oncology ( Site 1557), Rosario, Santa Fe Province
  - Centro de Urología (CDU) ( Site 1552), Buenos Aires
- Australia (4):
  - Macquarie University-MQ Health Clinical Trials Unit ( Site 1259), Macquarie University, New South Wales
  - Mater Hospital Brisbane ( Site 1257), South Brisbane, Queensland
  - Lyell McEwin Hospital ( Site 1252), Elizabeth Vale, South Australia
  - Frankston Hospital-Oncology and Haematology ( Site 1258), Frankston, Victoria
- Bulgaria (4):
  - MHAT "Uni Hospital" OOD ( Site 1154), Panagyurishte, Pazardzhik
  - Complex Oncology Center Plovdiv ( Site 1151), Plovdiv
  - MHAT Central Onco Hospital OOD ( Site 1158), Plovdiv
  - MHAT Serdika ( Site 1152), Sofia
- Canada (5):
  - BC Cancer - Vancouver Center ( Site 0110), Vancouver, British Columbia
  - CancerCare Manitoba ( Site 0108), Winnipeg, Manitoba
  - Moncton Hospital ( Site 0107), Moncton, New Brunswick
  - Ottawa Hospital Research Institute ( Site 0109), Ottawa, Ontario
  - Jewish General Hospital ( Site 0106), Montreal, Quebec
- China (7):
  - SUN YAT-SEN UNIVERSITY CANCER CENTRE ( Site 1406), Guangzhou, Guangdong
  - Sun Yat-sen Memorial Hospital, Sun Yat-sen University ( Site 1413), Guangzhou, Guangdong
  - Hunan Cancer Hospital ( Site 1403), Changsha, Hunan
  - Nanjing Drum Tower Hospital The Affiliated Hospital of Nanjing University Medical School-Urology ( Site 1404), Nanjing, Jiangsu
  - Nantong Tumor Hospital-Urology ( Site 1405), Nantong, Jiangsu
  - Fudan University Shanghai Cancer Center-Urology department ( Site 1401), Shanghai, Shanghai Municipality
  - Renji Hospital Shanghai Jiao Tong University School of Medicine ( Site 1402), Shanghai, Shanghai Municipality
- Colombia (5):
  - Fundacion Colombiana de Cancerología Clinica Vida ( Site 1653), Medellín, Antioquia
  - Clinica Colsanitas S.A, Sede Clínica Universitaria Colombia-Center Investigator ( Site 1654), Bogotá, Bogota D.C.
  - IMAT S.A.S ( Site 1652), Montería, Departamento de Córdoba
  - Fundación Cardiovascular de Colombia-Santander ( Site 1657), Piedecuesta, Santander Department
  - Fundación Valle del Lili ( Site 1656), Cali, Valle del Cauca Department
- Croatia (4):
  - Klinički bolnički centar Sestre milosrdnice ( Site 1703), Zagreb, City of Zagreb
  - Klinički bolnički centar Zagreb-Klinika za onkologiju ( Site 1701), Zagreb, City of Zagreb
  - Klinički bolnički centar Osijek ( Site 1705), Osijek, County of Osijek-Baranja
  - Klinički Bolnički Centar Split-Oncology and Radiotherapy ( Site 1702), Split, Split-Dalmatia County
- Czechia (4):
  - Fakultni nemocnice u sv. Anny v Brne ( Site 0253), Brno, South Moravian
  - Fakultni nemocnice Hradec Kralove-Klinika onkologie a radioterapie ( Site 0254), Hradec Králové
  - Fakultni Nemocnice Olomouc ( Site 0251), Olomouc
  - Fakultni Thomayerova nemocnice ( Site 0252), Prague
- France (10):
  - CHU La Timone ( Site 0456), Marseille, Bouches-du-Rhone
  - CHU Jean Minjoz ( Site 0453), Besançon, Doubs
  - C.H. regional Unv. de Brest - Hopital La Cavale Blanche - Institut de Cancerologie et d Imagerie ( Site 0461), Brest, Finistere
  - Institut Universitaire du Cancer Toulouse - Oncopole ( Site 0455), Toulouse, Haute-Garonne
  - CHU Limoges Hopital Dupuytren ( Site 0459), Limoges, Haute-Vienne
  - CHU GRENOBLE ALPES ( Site 0468), La Tronche, Isere
  - Centre Hospitalier Regional du Orleans ( Site 0463), Orléans, Loiret
  - Polyclinique du Bois ( Site 0458), Lille, Nord
  - Hopital Diaconesses Croix Saint Simon ( Site 0465), Paris
  - Gustave Roussy ( Site 0467), Villejuif, Île-de-France Region
- Germany (9):
  - Universitaetsklinikum Freiburg ( Site 0512), Freiburg im Breisgau, Baden-Wurttemberg
  - Universitaetsklinik fuer Urologie ( Site 0501), Tübingen, Baden-Wurttemberg
  - Caritas Krankenhaus St. Josef ( Site 0502), Regensburg, Bavaria
  - Universitaetsklinikum Wuerzburg ( Site 0520), Würzburg, Bavaria
  - Kath. Krankenhaus Marienhospital. Universitaetsklinik ( Site 0511), Herne, North Rhine-Westphalia
  - Universitaetsklinikum Muenster ( Site 0516), Münster, North Rhine-Westphalia
  - Universitaetsklinikum Carl Gustav Carus ( Site 0509), Dresden, Saxony
  - Krankenhaus Martha Maria Halle-Doelau ( Site 0507), Halle, Saxony-Anhalt
  - Vivantes Klinikum Am Urban ( Site 0519), Berlin
- Greece (5):
  - UNIVERSITY HOSPITAL OF PATRAS-DIVISION OF ONCOLOGY ( Site 0305), Pátrai, Achaia
  - General Hospital of Athens "Alexandra" ( Site 0303), Athens, Attica
  - Athens Medical Center ( Site 0304), Athens, Attica
  - ATTIKON GENERAL UNIVERSITY HOSPITAL ( Site 0301), Chaïdári, Attica
  - University General Hospital of Larissa ( Site 0302), Larissa, Thessaly
- Hungary (3):
  - Szegedi Tudományegyetem Szent-Györgyi Albert Klinikai Központ ( Site 1010), Szeged, Csongrád megye
  - Jász-Nagykun-Szolnok Vármegyei Hetényi Géza Kórház ( Site 1002), Szolnok, Jász-Nagykun-Szolnok
  - Debreceni Egyetem Klinikai Kozpont ( Site 1006), Debrecen
- Israel (7):
  - Rambam Health Care Campus-Oncology ( Site 0751), Haifa
  - Hadassah Medical Center-Oncology ( Site 0757), Jerusalem
  - Meir Medical Center-oncology ( Site 0754), Kfar Saba
  - Rabin Medical Center-Oncology ( Site 0752), Petah Tikva
  - Sheba Medical Center-ONCOLOGY ( Site 0753), Ramat Gan
  - Sourasky Medical Center-Oncology ( Site 0755), Tel Aviv
  - Yitzhak Shamir Medical Center-Oncology ( Site 0756), Ẕerifin
- Italy (8):
  - Fondazione IRCCS Istituto Nazionale dei Tumori-Struttura Complessa Oncologia Medica 1 ( Site 0588), Milan, Lombardy
  - Presidio Ospedaliero Santa Maria delle Grazie ( Site 0599), Pozzuoli, Napoli
  - AOU San Luigi Gonzaga di Orbassano ( Site 0595), Orbassano, Torino
  - Azienda Ospedaliera Universitaria Integrata Verona - Ospedale Borgo Trento ( Site 0598), Verona, Veneto
  - Azienda Ospedaliero Universitaria delle Marche-Clinica Oncologica ( Site 0593), Ancona
  - Ospedale Cannizzaro ( Site 0590), Catania
  - IRCCS Ospedale San Raffaele ( Site 0596), Milan
  - Istituto Oncologico Veneto IRCCS-Oncologia Medica 1 ( Site 0600), Padua
- Japan (17):
  - Nagoya University Hospital ( Site 1512), Nagoya, Aichi-ken
  - Hirosaki University Hospital ( Site 1501), Hirosaki, Aomori
  - University of Tsukuba Hospital ( Site 1502), Tsukuba, Ibaraki
  - Kanazawa University Hospital ( Site 1509), Kanazawa, Ishikawa-ken
  - Kitasato University Hospital ( Site 1506), Sagamihara, Kanagawa
  - Yokohama City University Medical Center ( Site 1508), Yokohama, Kanagawa
  - Kanagawa Cancer Center ( Site 1507), Yokohama, Kanagawa
  - Tohoku University Hospital ( Site 1503), Sendai, Miyagi
  - Hamamatsu University Hospital ( Site 1511), Hamamatsu, Shizuoka
  - Gifu University Hospital ( Site 1513), Gifu
  - Nagasaki University Hospital ( Site 1517), Nagasaki
  - Okayama University Hospital ( Site 1516), Okayama
  - Osaka International Cancer Institute ( Site 1514), Osaka
  - Osaka Metropolitan University Hospital ( Site 1515), Osaka
  - Institute of Science Tokyo Hospital ( Site 1505), Tokyo
  - Keio University Hospital ( Site 1504), Tokyo
  - Toyama University Hospital ( Site 1510), Toyama
- Malaysia (4):
  - University Malaya Medical Centre ( Site 0352), Lembah Pantai, Kuala Lumpur
  - Hospital Pulau Pinang ( Site 0355), George Town, Pulau Pinang
  - Sarawak General Hospital ( Site 0351), Kuching, Sarawak
  - Sunway Medical Centre ( Site 0353), Petaling Jaya, Selangor
- THE MEDICAL CITY ILOILO-The Medical City Iloilo - Clinical and Translational Research Institute-Ilo ( Site 0801), Iloilo City, Iloilo, Philippines
- Poland (6):
  - Clinical Research Center Medic-R ( Site 1061), Poznan, Greater Poland Voivodeship
  - Mazowiecki Szpital Wojewódzki w Siedlcach-Siedleckie Centrum Onkologii ( Site 1057), Siedlce, Masovian Voivodeship
  - Narodowy Instytut Onkologii ( Site 1051), Warsaw, Masovian Voivodeship
  - Wojewodzki Szpital im. Sw. Ojca Pio w Przemyslu ( Site 1053), Przemyśl, Podkarpackie Voivodeship
  - Uniwersytecki Szpital Kliniczny im. Jana Mikulicza-Radeckiego we Wrocławiu ( Site 1058), Wrocław, Silesian Voivodeship
  - Szpital Wojewodzki im. Mikolaja Kopernika ( Site 1055), Koszalin, West Pomeranian Voivodeship
- Portugal (4):
  - Unidade Local de Saude de Coimbra - Hospitais da Universidade de Coimbra ( Site 0406), Coimbra
  - Inst. Portugues de Oncologia de Lisboa Francisco Gentil EPE ( Site 0409), Lisbon
  - Unidade Local de Saude Lisboa Ocidental - Hospital de São Francisco Xavier ( Site 0401), Lisbon
  - Unidade Local de Saude de Santo António - Hospital Santo António ( Site 0408), Porto
- Romania (8):
  - MEMORIAL HEALTHCARE INTERNATIONAL S.R.L. ( Site 1104), Bucharest, București
  - Cardiomed SRL Cluj-Napoca ( Site 1101), Cluj-Napoca, Cluj
  - Institutul Oncologic Prof.Dr. Ion Chiricuta Cluj-Napoca ( Site 1102), Cluj-Napoca, Cluj
  - Institutul Oncologic Prof.Dr. Ion Chiricuta Cluj-Napoca ( Site 1103), Cluj-Napoca, Cluj
  - SC Radiotherapy Center Cluj SRL ( Site 1108), Comuna Floresti, Cluj
  - S.C. Centrul de Oncologie Sf. Nectarie SRL ( Site 1107), Craiova, Dolj
  - Policlinica Oncomed SRL ( Site 1106), Timișoara, Timiș County
  - Institutul Oncologic Cluj-Oncologie Medicala ( Site 1109), Cluj-Napoca
- Russia (11):
  - Altay Regional Oncology Dispensary ( Site 0851), Barnaul, Altayskiy Kray
  - National Medical Research Radiology Centre ( Site 0869), Obninsk, Kaluzskaja Oblast
  - National Medical Research Centre of Oncology named after N.N. Blokhin ( Site 0865), Moscow, Moscow
  - First Moscow State Medical University n.a. I.M.Sechenov ( Site 0871), Moscow, Moscow
  - Volga District Medical Center ( Site 0876), Nizhny Novgorod, Nizhny Novgorod Oblast
  - St.Petersburg Clinical Hospital RAS ( Site 0864), Saint Petersburg, Sankt-Peterburg
  - St.Petersburg State Medical Univ. n.a. acad. I.P.Pavlov ( Site 0856), Saint Petersburg, Sankt-Peterburg
  - Scientific Research Oncology Institute n.a. N.N.Petrov ( Site 0852), Saint Petersburg, Sankt-Peterburg
  - Sverdlovsk Regional Oncology Hospital ( Site 0867), Yekaterinburg, Sverdlovsk Oblast
  - Sverdlovsky Regional Clinical hospital #1 ( Site 0868), Yekaterinburg, Sverdlovsk Oblast
  - Volgograd Regional Uronephrological Center ( Site 0870), Volzhsky, Volgograd Oblast
- Tan Tock Seng Hospital ( Site 0704), Singapore, Central Singapore, Singapore
- South Africa (3):
  - Wits Clinical Research ( Site 0603), Johannesburg, Gauteng
  - Steve Biko Academic Hospital ( Site 0601), Pretoria, Gauteng
  - Groote Schuur Hospital ( Site 0602), Cape Town, Western Cape
- South Korea (7):
  - Chonnam National University Hwasun Hospital ( Site 1353), Jeollanam-do, Jeonranamdo
  - Seoul National University Bundang Hospital ( Site 1355), Gyeonggi-do, Kyonggi-do
  - Kyungpook National University Chilgok Hospital ( Site 1354), Daegu, Kyongsangbuk-do
  - Asan Medical Center ( Site 1352), Songpagu, Seoul
  - Gachon University Gil Medical Center ( Site 1356), Incheon
  - Korea University Anam Hospital ( Site 1357), Seoul
  - Seoul National University Hospital ( Site 1351), Seoul
- Spain (10):
  - Hospital Germans Trias i Pujol. ICO de Badalona ( Site 0658), Badalona, Barcelona
  - Xarxa Assistencial Universitaria Manresa ( Site 0655), Manresa, Barcelona
  - Institut Català d'Oncologia (ICO) - Girona ( Site 0653), Girona, Gerona
  - CHUS - Hospital Clinico Universitario-Servicio de Oncologia ( Site 0660), Santiago de Compostela, La Coruna
  - Hospital Universitario Insular de Gran Canaria ( Site 0657), Las Palmas de Gran Canaria, Las Palmas
  - Hospital Universitario Central de Asturias ( Site 0654), Oviedo, Principality of Asturias
  - Fundación Instituto Valenciano de Oncología-Oncologico ( Site 0662), Valencia, Valenciana, Comunitat
  - Hospital Universitari Vall d'Hebron-Departamento de Oncologia- VHIO ( Site 0661), Barcelona
  - Hospital Clinico Universitario San Carlos de Madrid ( Site 0651), Madrid
  - Hospital Virgen del Rocio ( Site 0659), Seville
- Taiwan (3):
  - Chang Gung Memorial Hospital at Kaohsiung ( Site 1203), Kaohsiung City
  - China Medical University Hospital ( Site 1202), Taichung
  - Taipei Veterans General Hospital ( Site 1201), Taipei
- Ukraine (7):
  - I.I. Mechnykov Dnipropetrovsk Regional Clinical Hospital ( Site 0959), Dnipro, Dnipropetrovsk Oblast
  - MI Clinical oncology dispensary of Dnipropetrovsk regional council ( Site 0954), Dnipro, Dnipropetrovsk Oblast
  - Regional Clinical Center of Urology and Nephrology n.a. V.I. Shapoval ( Site 0952), Kharkiv, Kharkivs’ka Oblast’
  - MNPE Regional Center of Oncology ( Site 0955), Kharkiv, Kharkivs’ka Oblast’
  - Municipal Non-profit Enterprise of Kharkiv Regional Council RCSDRPP ( Site 0965), Kharkiv, Kharkivs’ka Oblast’
  - Lviv Oncology Regional Treatment and Diagnostic Center ( Site 0960), Lviv, Lviv Oblast
  - Zhytomyr Regional Oncology Center ( Site 0961), Zhytomyr, Zhytomyr Oblast
- United Kingdom (3):
  - Torbay Hospital ( Site 1804), Torquay, Devon
  - Charing Cross Hospital-Oncology Research ( Site 1802), London, Hammersmith and Fulham
  - St Bartholomew's Hospital-Centre for Experimental Cancer Medicine ( Site 1801), London, London, City of

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26290&tenant=MT_MSD_9011